CLINICAL TRIAL: NCT06667557
Title: Comparison of Super Pulse Fiber Thulium Laser and Holmium Laser Lithotripsy Under Ureteroscopy
Brief Title: Comparing Super Pulse Fiber Thulium Laser and Holmium Laser for Ureteral Stone Fragmentation During Ureteroscopy
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yi Shao, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: IIT2024-147
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Kidney Calculi
MeSH Terms: conditions — Kidney Calculi | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sTFL Group: Kidney stones and/or upper ureteral stones are treated with a superpulsed thulium fiber laser (sTFL)
  Interventions: Device: Superpulse Thulium Fiber Laser (sTFL) Treatment
- Ho:YAG Group: Kidney stones and/or upper ureteral stones are treated with a holmium :YAG laser (Ho:YAG)
  Interventions: Device: Holmium:YAG Laser (Ho:YAG) Treatment

INTERVENTIONS:
Device: Superpulse Thulium Fiber Laser (sTFL) Treatment — The superpulse thulium fiber laser (sTFL) was used as a minimally invasive surgical treatment for kidney and upper ureteral stones. All procedures were performed by experienced urologists using standard techniques for laser lithotripsy. Laser settings, such as pulse energy and frequency, were adjusted according to stone characteristics and the surgeon's judgment to optimize treatment efficacy and safety.
  Groups: sTFL Group
Device: Holmium:YAG Laser (Ho:YAG) Treatment — The holmium:YAG laser (Ho:YAG) was used as a minimally invasive surgical treatment for kidney and upper ureteral stones. All procedures were performed by experienced urologists using standard techniques for laser lithotripsy. Laser settings, such as pulse energy and frequency, were adjusted according to stone characteristics and the surgeon's judgment to optimize treatment efficacy and safety.
  Groups: Ho:YAG Group

SUMMARY:
The goal of this prospective, multicenter, randomized controlled trial is to objectively evaluate the clinical efficacy and safety differences between superpulse thulium fiber laser (sTFL) and holmium:YAG laser (Ho:YAG) in flexible ureteroscopy (FURS) lithotripsy in adult patients aged 18-70 years with kidney stones and/or upper ureteral stones (6-20mm). The main questions it aims to answer are:

Does sTFL yield a higher stone-free rate (SFR) compared to Ho:YAG at 3 months post-FURS? Is sTFL superior to Ho:YAG in terms of operation time, complication rate, and surgeon's visual experience during FURS? Researchers will compare the experimental group receiving sTFL treatment to the control group receiving Ho:YAG laser treatment to see if sTFL demonstrates better lithotripsy efficiency, safety, and ease of operation.

Participants aged 18-70 years will:

Undergo FURS lithotripsy under general anesthesia using either sTFL (experimental group) or Ho:YAG laser (control group) based on randomization Have CT scans at 3 months post-operation to assess stone-free status Be monitored for intraoperative and postoperative complications Have surgeons rate their visual experience during the procedure in terms of visual clarity, lithotripsy efficiency, stone movement and tissue injury

DETAILED DESCRIPTION:
Flexible ureteroscopy (FURS) has become a widely accepted minimally invasive treatment modality for kidney stones and upper ureteral stones. Holmium:YAG laser (Ho:YAG) is currently the gold standard for laser lithotripsy during FURS. However, the superpulse thulium fiber laser (sTFL) has emerged as a promising alternative with potential advantages in terms of lithotripsy efficiency and safety. This prospective, multicenter, randomized controlled trial aims to objectively evaluate the clinical efficacy and safety differences between sTFL and Ho:YAG in FURS for adult patients with kidney stones and/or upper ureteral stones (6-20mm).

The study will enroll 136 participants aged 18-70 years with confirmed diagnosis of kidney stones and/or upper ureteral stones (6-20mm) based on CT scans. Participants will be randomized in a 1:1 ratio to undergo FURS with either sTFL (experimental group) or Ho:YAG (control group). The primary outcome measure will be the stone-free rate (SFR) at 3 months post-operation, defined as residual fragments <2mm on CT scans. Secondary outcomes will include operation time, intraoperative complications (e.g., ureteral injury, bleeding, infection), postoperative complications (e.g., fever, hematuria), changes in vital signs, surgeon's visual experience, and stone recurrence rate at 6 months.

Participants will be closely monitored for adverse events and complications throughout the study period. The Clavien-Dindo classification system will be used to grade postoperative complications. Detailed safety assessments will be performed, including recording of adverse events, reporting of serious adverse events, monitoring of vital signs, and evaluation of complications.

The study will consist of the following visits:

Baseline visit (screening period): Participants will provide informed consent, undergo eligibility assessment, and have their demographic information, medical history, vital signs, and CT scans collected.

Intraoperative visit (treatment period): Researchers will record operation time, laser type used, surgeon's visual experience, and monitor vital signs and complications.

Postoperative visits (treatment period): Participants will be closely monitored for vital signs, symptoms, and complications within 24 hours after surgery.

Follow-up visits at 3 months and 6 months (follow-up period): Participants will undergo CT scans to assess stone clearance and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Diagnosis of kidney stones and/or upper ureteral stones with stone diameter ≥6mm and ≤20mm
* Plan to undergo fURS lithotripsy
* General anesthesia to complete the operation
* The latest urine culture before surgery is negative
* Signed and dated informed consent indicating that the patient or his or her legal representative has been fully informed about the study and has consented to participate

Exclusion Criteria:

* Isolated kidney
* Previous history of kidney transplantation or urinary diversion surgery
* Congenital malformations of urinary system
* Abnormal coagulation mechanism due to blood system diseases, liver diseases, etc.
* Severe heart or lung disease, malignancy and immune deficiency status
* Neurogenic bladder
* Failure to provide informed consent
* Have an untreated urinary tract infection
* The presence of known anatomic abnormalities (such as ureteral stenosis), urothelial tumors, or stones that can be removed directly without the use of laser lithotripsy
* Pregnant women
* In cases where the stone cannot be reached with a bendable negative pressure suction sheath, or in cases where the stone cannot be reached with a conventional sheath or the pyeloureteral junction
* Surgical completion under epidural anesthesia or lumbar anesthesia
* Recurrent stones due to genetic metabolic diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-70 years who plan to undergo fURS lithotripsy for kidney stones and/or upper ureteral stones (6-20mm)
Sampling Method: Non-Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-10-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Stone-free Rate | 3 months post-procedure
  The proportion of participants achieving complete stone clearance, defined as no residual fragments or residual fragments ≤2 mm on follow-up imaging (e.g., plain radiography, ultrasound, or computed tomography) after a single laser lithotripsy procedure.

SECONDARY OUTCOMES:
Operative Time | Measured during the procedure
  The duration of the surgical procedure, measured in minutes from the start of the operation until the completion of the surgical procedure. Operative times will be recorded and compared between the two groups.
Complication Rate | From the start of the procedure until 24 hours post-procedure
  The proportion of participants experiencing complications during the surgical procedure and within 24 hours after the procedure. Complications will be recorded and classified according to the Clavien-Dindo system, which categorizes surgical complications by severity. The complication rates will be compared between the two groups.
Surgeon's Visual Experience | Measured immediately after the procedure
  The surgeon's subjective assessment of visual clarity, stone fragmentation efficiency, stone movement, and tissue damage during the procedure. Recording the subjective feelings of urologists.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Shao, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No